CLINICAL TRIAL: NCT06438380
Title: Experience of Critically Ill Patients in the Use of a Telemedicine Platform for the Follow-up of Post Intensive Care Syndrome (PICS) After ICU Discharge
Brief Title: User Experience of a Telemedicine Platform for the Follow-up of Post Intensive Care Syndrome (PICS)
Status: Not yet recruiting | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/5126
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Critical Illness
Keywords: Qualitative research; Post-Intensive Care Syndrome
MeSH Terms: conditions — Critical Illness; postintensive care syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Survivors of critical illness may present with a set of physical, emotional and cognitive sequelae, known as Post Intensive Care Syndrome (PICS). These alterations can become chronic over time and significantly affect patients' quality of life. Therefore, follow-up and monitoring of critically ill patients after ICU discharge, for example through telemedicine, could be essential for the prevention, early detection and management of PICS.

Our main objective is to evaluate the suitability and user experience of a telemedicine platform from the perspective of critically ill patients. This study proposes the participation of ICU survivors in the design and improvement of a telemedicine platform for PICS follow-up through a qualitative approach. Participants will test the platform in person three months after discharge from the ICU and then undergo a semi-structured interview to assess their experience. The findings derived from this study may contribute to improve both the content and the format of the platform, optimizing resources and facilitating the management of post-ICU sequelae, which will have a positive impact on the patient's recovery process.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years)
* Admitted to a medical/surgical ICU
* For respiratory failure, cardiogenic shock, or septic shock
* With an expected ICU stay of ≥48 hours
* Catalan and/or Spanish speakers
* Who are able to give informed consent by themselves

Exclusion Criteria:

* History of intellectual disability or other neurodevelopmental disorders, such as autism spectrum disorder
* History of neurological disorders, dementia or other neurodegenerative diseases, such as epilepsy, Alzheimer's disease, Parkinson's disease or multiple sclerosis
* History of brain damage, such as traumatic brain injury or stroke
* History of severe psychiatric illness, such as psychotic, bipolar, depressive, obsessive-compulsive, post-traumatic or personality disorder
* Suspected or confirmed substance use disorder
* Suspected or confirmed communicable disease in an isolated patient
* Uncorrected hearing or visual impairment
* Enrolled in another trial that does not allow co-enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted to the ICU of the Parc Tauli Hospital (Sabadell, Spain).
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
1:1 semi-structured interviews | 3 months after ICU discharge
  To evaluate the user experience of a telemedicine platform for monitoring post-intensive care syndrome from the perspective of critically ill patients after ICU discharge through semi-structured interviews